CLINICAL TRIAL: NCT03749551
Title: TowaRds Understanding the phEnoTYPEs of Cardiovascular Dysfunction in Patients With Chronic Kidney Disease and HaemoDialysis Using Cardiovascular Magnetic Resonance Imaging - TRUE-Type-CKD Study
Brief Title: Towards Understanding the Phenotype of Cardiovascular Disease in CKD - TRUE-Type-CKD Study
Acronym: TRUE-TypeCKD
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Valentina Puentmann, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: TrueTypeCKD 4/17
Record Dates: First submitted 2018-11-17; First posted 2018-11-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Cardiomyopathies; Chronic Kidney Diseases; Hypertrophy, Left Ventricular
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Renal Insufficiency, Chronic; Hypertrophy, Left Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: diagnostic test - patients serving as their own controls
  Interventions: Diagnostic Test: cardiac magnetic resonance (CMR) post haemodialysis

INTERVENTIONS:
Diagnostic Test: cardiac magnetic resonance (CMR) post haemodialysis — patients will undergo a second CMR scan immediately after receiving haemodialysis (native CMR study)

SUMMARY:
Premature cardiovascular disease (CVD) is the leading cause of death in patients with kidney disease (CKD). Excessive cardiac mortality is thought to be secondary to non-atherosclerotic processes, with left ventricular (LV) hypertrophy (LVH) and remodelling being the predominant phenotypical features. Along with other risk factors, subclinical ischaemia and haemodynamic perturbations associated with haemodialysis (HD) are thought to contribute to the ultimate development of LV systolic and diastolic dysfunction. The development of these adverse features reflects a specific cardiomyopathy due to CKD and subsequently, to uraemia. Patients receiving hemodialysis (HD) have a higher incidence rate of heart failure (predominantly with preserved ejection fraction), with phenotypically eccentric hypertrophic remodelling, systolic and diastolic dysfunction as well as high rate of interstitial myocardial fibrosis. Detection and ultimately reversal of the development of this CKD-related cardiomyopathy are important goals for improving the CVD, morbidity and mortality of CKD patients.The objectives of this study are, firstly, to investigate the complex myocardial phenotype in patients with various stages of CKD, secondly, to relate the CMR-measures to outcome, and thirdly, to be able to estimate the effects of chronic uremia/hypervolemia. Deciphering the predominant driver of remodelling on an individual level may help to personalise anti-remodelling strategies. Native T1 and T2 mapping imaging provide non-invasive imaging tools to detect myocardial fibrosis and oedema, respectively. Prognostic associations of these measures may clarify the relative prevalence of adverse phenotype and their relative contribution to adverse events and poor outcome. The role of chronic water retention and uraemia may be associated with interstitial myocardial oedema promoting further the remodelling process.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >18 years of age
2. Able to provide informed consent
3. Chronic kidney disease stages G3-5 (eGFR<59 ml/min/1.73m2)

Exclusion Criteria:

1. Absence of absolute clinical indication for MRI studies (MR unsafe or incompatible devices, aneurysm clips, cochlear implants, loose metal foreign objects)
2. Absolute contraindications to gadolinium contrast agent (previous allergic reaction or pregnancy),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with established diagnosis of chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
survival | 1 year
  number of deaths
survival | 5 year
  number of deaths
rate of death due to cardiovascular causes | 1 year
  number of participants died due to death due to myocardial infarction, sudden cardiac death, heart failure
rate of death due to cardiovascular causes | 5 year
  number of participants died due to death due to myocardial infarction, sudden cardiac death, heart failure

SECONDARY OUTCOMES:
rate of heart failure events | 1 year
  number of participants with heart failure death and hospitalisation due to heart failure
rate of heart failure events | 5 year
  number of participants with heart failure death and hospitalisation due to heart failure

OTHER OUTCOMES:
Change in native T1 and T2 (in msec) pre and post haemodialysis | 24 hour
  measurement of change in magnetisation relaxation (in msec)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arcari L, Engel J, Freiwald T, Zhou H, Zainal H, Gawor M, Buettner S, Geiger H, Hauser I, Nagel E, Puntmann VO. Cardiac biomarkers in chronic kidney disease are independently associated with myocardial edema and diffuse fibrosis by cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2021 Jun 7;23(1):71. doi: 10.1186/s12968-021-00762-z. PMID 34092229
- [Result] Valbuena-Lopez SC, Camastra G, Cacciotti L, Nagel E, Puntmann VO, Arcari L. Cardiac Imaging Biomarkers in Chronic Kidney Disease. Biomolecules. 2023 Apr 29;13(5):773. doi: 10.3390/biom13050773. PMID 37238643
- [Result] Chen M, Arcari L, Engel J, Freiwald T, Platschek S, Zhou H, Zainal H, Buettner S, Zeiher AM, Geiger H, Hauser I, Nagel E, Puntmann VO. Aortic stiffness is independently associated with interstitial myocardial fibrosis by native T1 and accelerated in the presence of chronic kidney disease. Int J Cardiol Heart Vasc. 2019 Jun 26;24:100389. doi: 10.1016/j.ijcha.2019.100389. eCollection 2019 Sep. PMID 31304234
- [Result] Arcari L, Hinojar R, Engel J, Freiwald T, Platschek S, Zainal H, Zhou H, Vasquez M, Keller T, Rolf A, Geiger H, Hauser I, Vogl TJ, Zeiher AM, Volpe M, Nagel E, Puntmann VO. Native T1 and T2 provide distinctive signatures in hypertrophic cardiac conditions - Comparison of uremic, hypertensive and hypertrophic cardiomyopathy. Int J Cardiol. 2020 May 1;306:102-108. doi: 10.1016/j.ijcard.2020.03.002. Epub 2020 Mar 3. PMID 32169347